CLINICAL TRIAL: NCT06152484
Title: A Study on Evaluating the Consistency of CASIA2, Pentacam, and Corvis ST Measurement Parameters and the Diagnostic Efficacy of Early Keratoconus
Brief Title: Evolution of a Novel Optical Coherence Tomography Based Index in Diagnosing Keratoconus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023063
Record Dates: First submitted 2023-10-30; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Scansys, Pentacam, Keratoconus, Subclinical Keratoconus
Keywords: Scansys, Pentacam, Keratoconus, subclinical keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normal control group
  Interventions: Other: Pentacam, Corvis ST and CASIA2
- Subclinical keratoconus
  Interventions: Other: Pentacam, Corvis ST and CASIA2
- Keratoconus
  Interventions: Other: Pentacam, Corvis ST and CASIA2

INTERVENTIONS:
Other: Pentacam, Corvis ST and CASIA2 — morphological and biomechanical parameters of corneal were obtain by CASIA2, Pentacam and Corvis ST

SUMMARY:
Comparison of corneal topography based on oct OCT principle (CASIA2) with Pentacam and Scheimpflug-based biomechanical devices (Corvis ST) in screening and diagnosing keratoconus; and evaluation of the consistency with Pentacam in measuring corneal parameters (such as curvature and thickness).

ELIGIBILITY:
Inclusion Criteria:

1. Best corrected visual acuity (BCVA) ≥ 20/20;
2. No other eye diseases except myopia and astigmatism;
3. The cornea was transparent, and there was no cloud or pannus;

Exclusion Criteria:

1. The presence of ocular diseases other than myopia and keratoconus;
2. Ocular trauma;
3. Previous ocular surgery; 4 Patients were required to stop wearing soft contact lenses for at least 2 weeks and rigid contact lenses for at least 4 weeks before examination; 6. Pregnant and lactating women;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients premedicated for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
screening and diagnosis ability | one year
  Evaluate the sensitivity and specificity of parameters measured by CASIA2, Pentacam in diagnosing keratoconus using Receiver operating characteristic curves (ROC), and compare the Ectasia Screening Similarity（ESS）and D-value diagnostic efficacy using Area under the ROC curve (AUROC). Use the Delong test to compare the accuracy of various parameters in diagnosing early keratoconus.

SECONDARY OUTCOMES:
Measurement consistency | one year
  The independent sample T-test is used to compare inter- group differences in baseline data. Use independent sample T-test and One-way ANOVA to evaluate the consistency of the measurement results (anterior and posterior corneal curvature, corneal refractive index, CCT) obtained by CASIA2 and Pentacam.Finally, the ultimate outcome（such ad：K1 K2 KMax CCT） indicates that the P-value between the two devices is less than 0.05 and ICC-value is more than 0.75.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tiajin Eye Hospita
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided